CLINICAL TRIAL: NCT04788823
Title: The Impact of Prednisone on Semen Parameters and Pregnancy Rates Post Vasectomy Reversal: A Randomized, Controlled Trial
Brief Title: The Impact of Prednisone on Semen Parameters and Pregnancy Rates Post Vasectomy Reversal
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Charitable Union for the Research and Education of Peyronie's Disease (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUREPD 102
Record Dates: First submitted 2021-03-03; First posted 2021-03-09 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Vasectomy Reversal
MeSH Terms: interventions — Prednisone

STUDY DESIGN:
Intervention Model Description: The study cohort will be randomized to one of 4 arms: control or 3 different drug protocols.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control (No Intervention): Group 1 will represent controls and will not receive prednisone in the 3-year post-op period.
- Prednisone Monthly - Scheduled (Experimental): Group 2 will receive 3, one-month courses of prednisone (20 mg daily x 1 week, 10 mg daily x 1 week, 5 mg x 2 weeks). These will be given at the beginning of months 0, 2, and 4 and will be self-administered.
  Interventions: Drug: Prednisone
- Prednisone Monthly - As Needed (Experimental): Group 3 will receive a maximum of 3, one-month courses of prednisone (20 mg daily x 1 week, 10 mg daily x 1 week, 5 mg x 2 weeks). These will be administered based on sequential semen analyses. If a semen analysis demonstrates a drop in concentration from a prior analysis or if it shows a 0 concentration, the course will be administered.
  Interventions: Drug: Prednisone
- Prednisone Every Other Week (Experimental): Group 4 will receive alternating 1 week dosages of prednisone (1 week on, 1 week off - 5 mg daily only) for a total of 24 weeks
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Prednisone — Treatment groups will be administered different dosages of Prednisone post vasectomy reversal.
  Arms: Prednisone Every Other Week; Prednisone Monthly - As Needed; Prednisone Monthly - Scheduled

SUMMARY:
1. Determine impact of prednisone on semen parameters post vasectomy reversal (evaluated both using prednisone as a combined cohort as well as via 3 separate protocols).
2. Determine impact of prednisone on pregnancy rates post vasectomy reversal (evaluated both using prednisone as a combined cohort as well as via 3 separate protocols).
3. Assess adverse events with prednisone utilization

DETAILED DESCRIPTION:
1. Introduction

This document is a protocol for a randomized, controlled clinical trial. This study will be carried out in accordance with the procedures described in this protocol, applicable United States government regulations and Western International Review Board policies and procedures.

1.1 Background and Clinical Need for the Current Study

Currently, vasectomy reversals are a common surgical treatment performed to restore fertility in men who have previously undergone vasectomies. Post-operatively, sperm are seen in the ejaculate in the majority of men undergoing a reversal, however, sperm counts commonly fluctuate over time. In a percentage of men, counts will ultimately decline to 0 over time. Although the exact cause of this decline is unknown, it is felt to be secondary to tissue remodeling and/or inflammation leading to stenosis of the anastomotic repair. To address this issue, clinicians have used prednisone for several decades. Despite the long-standing use, very few publications have assessed the overall efficacy of this therapy on improving outcomes. The objective of the current study is to perform a much more robust assessment as to the true risks and benefits of this therapy in improving post-operative outcomes.

1.2 Investigational Treatments

Men who are post vasectomy reversal will be treated with either no therapy (control) or one of three separate protocols with prednisone.

1.3 Preliminary Data

A very limited amount of data exists regarding the efficacy of corticosteroids in improving outcomes post vasectomy reversal. The earliest known study involved the use of cortisone in 8 dogs who underwent vasovasostomy procedures. Results showed that 63% of vasa were patent in the steroid group compared to 43% in control animals (not statistically significant). A second study administered prednisone to 20 men post vasectomy reversal and compared against 20 men who had previously undergone reversal but were not treated with prednisone. Results showed improved sperm counts (statistically significant) without statistically significant differences in pregnancy rates. And finally, a third study performed a retrospective analysis in 89 men who underwent reversals over a period of 11 years. Results demonstrated increases in total motile sperm counts, with greater improvements noted among men who exhibited the presence of sperm at the time of prednisone administration compared to those with 0 sperm.

These data are limited by several factors. The first study listed also performed a pathologic analysis and failed to demonstrate any differences in the extent of fibrosis. The second study was performed in a sequential manner, where outcomes may have just been reflective of learning curve improvements, and improvements were no longer present after the steroid was discontinued. The third study was retrospective in nature, and therefore is limited by significant biases (i.e. only men with low counts received the treatment, which leads to an effect bias). All series were very small and lacked statistical power.

Despite these limited data, the use of prednisone post vasectomy reversal is a common, widespread practice among reversal surgeons.

1.4 Study Rationale and Risk Analysis (Risks to Benefits Ratio)

The study is currently designed to address an important clinical question. Specifically, does the addition of prednisone post-operatively lead to improved semen and pregnancy outcomes. Additionally, does the addition of prednisone lead to temporary or permanent improvements. Regarding potential risks, the use of prednisone will be limited to shorter durations of therapy. Potential risks in a young, healthy population are low. Specifically, an analysis of men 20-64 found that the risks of prednisone include 3 GI bleeds per 100 person years, <1 with a severe infection, and <1 with heart failure. Our study will not include as high of a dosage or duration of therapy shown in this prior risk study, and as such, the true risks are anticipated to be small (if any).

ELIGIBILITY:
Inclusion Criteria:

* Men undergoing a first-time vasectomy reversal at the Male Fertility and Peyronie's Clinic
* 18-65 years of age
* Current sexual partner with desire to achieve pregnancy immediately
* Intent of reversal to restore fertility
* Partner <36 years of age
* Partner with no known fertility issues
* Prior history of paternity

Exclusion Criteria:

* Current corticosteroid use
* Prior vasectomy reversal
* Prior chemotherapy
* Testosterone use within 1 year of the vasectomy reversal
* Solitary testicle
* History of diabetes mellitus
* History of systemic fungal infection
* Hypertension
* Any degree of diagnosed renal insufficiency
* Partner on birth control within past 3 months

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-02-24 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Impact of Prednisone on semen concentration post vasectomy reversal | 3 years
  Determine impact of prednisone on semen concentration post vasectomy reversal (evaluated both using prednisone as a combined cohort as well as via 3 separate protocols).
Impact of prednisone on pregnancy rates post vasectomy reversal. | 3 Years
  Determine impact of prednisone on pregnancy rates post vasectomy reversal (evaluated both using prednisone as a combined cohort as well as via 3 separate protocols).
Assess adverse events with prednisone utilization | 3 years
  Assess adverse events with prednisone utilization

SECONDARY OUTCOMES:
Impact of Prednisone on semen concentration post vasectomy reversal | 1 year
  Determine impact of prednisone on semen concentration post vasectomy reversal (evaluated both using prednisone as a combined cohort as well as via 3 separate protocols).
Impact of prednisone on pregnancy rates post vasectomy reversal. | 1 year
  Determine impact of prednisone on pregnancy rates post vasectomy reversal (evaluated both using prednisone as a combined cohort as well as via 3 separate protocols).
Impact of Prednisone on semen concentration post vasectomy reversal | Up to 1 year
  Determine impact of prednisone on semen concentration post vasectomy reversal (evaluated both using prednisone as a combined cohort as well as via 3 separate protocols).

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Green, Study Director — The Male Fertility and Peyronie's Clinic
Locations (1):
- Cure PD, Orem, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trost L, Helo S, Brearton K, Warner R, Ziegelmann M, Kohler T, Savage J. Impact of prednisone on vasectomy reversal outcomes (iPRED study): results from a randomized, controlled clinical trial. Fertil Steril. 2025 May;123(5):804-811. doi: 10.1016/j.fertnstert.2024.11.019. Epub 2024 Nov 20. PMID 39577828